CLINICAL TRIAL: NCT02351453
Title: Patients With Alzheimer Disease, Spouse Carers and Risk of Institutionalization: a Prospective Observational Cohort Study of Dyads (AID Study)
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2011/24
Record Dates: First submitted 2015-01-13; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2011-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of AID study is to identify the medico-neuropsychological, socio-economic and environmental baseline characteristics of dyads associated with the institutionalization of AD patients.

DETAILED DESCRIPTION:
In order to reduce Alzheimer Disease (AD) adverse impacts at individual level as well as in terms of expenditures, the development of efficient strategies based on the identification and the correction of risk factors of institutionalization of AD patients proves necessary.

While it has been identified that institutionalization date depends on patients' health characteristics, the role of social, economic and environmental factors still remains few known.

The investigators hypothesized that institutionalization of AD patients could be related not only to medico-neuropsychological patients' characteristics but also to socio-economic and environmental characteristics of dyad (i.e., AD patient and spouse carer), that could modify the delay of institutionalization.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria for AD patients were:

  * Over age 65,
  * Diagnosis of AD according to the NINCDS-ADRDA ( National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association) criteria,
  * Last memory center consultation between 6 and 12 months before the inclusion,
  * Being affiliated to the French health insurance,
  * Living at home,
  * Having a caregiver with inclusion criteria,
  * Agreement of General Practitioner (GP) of AD patient to participate in the study and affiliation of the GP to the national "Association pour le Développement de l'Information Médicalisée" (ADIM) French network.
* Eligibility criteria for spouse carers were:

  * Over age 65,
  * Being the spouse and the caregiver of AD patient,
  * Being affiliated to the French health insurance,
  * Living at home with AD patient.

Exclusion Criteria:

* Non inclusion criteria for AD patients and spouse carers were:

  * An inability to understand and speak French,
  * Acute disease in the past month of baseline assessment,
  * Expected moving outside the recruitment area during the follow-up period
  * Concomitant participation in a clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: AD patients and their spouses were recruited in each memory clinic by a physician during the annual follow-up consultation of AD patient based on eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2011-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Date of institutionalization of AD patients (standardized questionnaire) | This outcome is assessed at 12 months.
  Date of entrance in institution was collected by a standardized questionnaire.

SECONDARY OUTCOMES:
The increase formal home help services (measured by a standardized questionnaire and coded as a binary variable) | This outcome is assessed at baseline and 12 months.
  The use of formal home help services was measured by a standardized questionnaire and coded as a binary variable.
The delay of institutionalization of AD patients (assessed by a standardized questionnaire and expressed in number of days) | This outcome is assessed at baseline and 12 months.
  The delay of institutionalization was assessed by a standardized questionnaire and expressed in number of days.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- University Hospital, Angers, France